CLINICAL TRIAL: NCT05340530
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of Injectable TQD3606 in a Single Center, Randomized, Double-blind, Placebo-controlled, Single, Multiple Dosing in Healthy Subjects, and to Explore Urinary Excretion of the Product
Brief Title: To Evaluate the Pharmacokinetic Effects of TQD3606 for Injection in Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: TQD3606-I-01
Record Dates: First submitted 2022-04-01; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Infections
MeSH Terms: conditions — Infections | interventions — Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- The injectable TQD3606 (Experimental): received a single dose of 0.75g TQD3606 for injection
  Interventions: Drug: The injectable TQD3606
- The injectable TQD3606+ meropenem (Active Comparator): First, a single dose of 0.5g of meropenem for injection was administered for 0.5h intravenous infusion; after washout for at least 2 days, 0.75g of TQD3606 for injection was administered for 1h intravenous infusion; for at least 2 days of washout, 0.75g was administered A single dose of TQD3606 for injection was administered for 2 hours, and the elution time was at least 2 days. Finally, a single dose of 0.75 g of TQD3606 for injection was administered, and the duration of intravenous infusion was 3 hours.
  Interventions: Drug: The injectable TQD3606; Drug: meropenem
- The injectable TQD3606+ meropenem+ Avibactam Sodium (Active Comparator): According to the random table, they were divided into two groups, A and B, Group A was given 1.0g meropenem for injection (Mepin) in the first cycle, and 0.5g avibactam sodium for injection in the second cycle. The third cycle was given 1.5g TQD3606 for injection; group B was given 0.5g avibactam sodium for injection in the first cycle, 1.0g meropenem (Mepin) for injection in the second cycle, and 1.5g for injection in the third cycle TQD3606.
  Interventions: Drug: The injectable TQD3606; Drug: meropenem; Drug: Avibactam Sodium
- The injectable TQD3606-1 (Experimental): First, 0.75g TQD3606 for injection was administered multiple times (Dosing every 8 hours, 3 consecutive doses), and at least 2 days were washed out after the last dose; then 1.125g TQD3606 for injection was administered multiple times (Dosing every 12 hours, 2 consecutive doses) times), wash out at least 2 days after the last administration; finally, a single administration of 2.25 g of TQD3606 for injection (Dosing every 12 hours, once administered). Intravenous infusion for 3 hours.
  Interventions: Drug: The injectable TQD3606
- The injectable TQD3606/ Placebo (Placebo Comparator): First, a single dose of 3.0g TQD3606 for injection/placebo was administered, intravenous infusion for 3hours, and washout for at least 3 days; then multiple doses of 3.0g TQD3606 for injection/placebo were administered (Dosing every 8 hours, 10 consecutive doses) , the intravenous infusion duration is 3hours.
  Interventions: Drug: The injectable TQD3606; Drug: Placebo

INTERVENTIONS:
Drug: The injectable TQD3606 — TQD3606 is a fixed-dose combination of meropenem and avibatam.
Drug: meropenem — Meropenem is a carbapenem antibiotic
  Arms: The injectable TQD3606+ meropenem; The injectable TQD3606+ meropenem+ Avibactam Sodium
Drug: Avibactam Sodium — Avibactam is beta-lactamase inhibitor.
  Arms: The injectable TQD3606+ meropenem+ Avibactam Sodium
Drug: Placebo — It is a placebo.
  Arms: The injectable TQD3606/ Placebo

SUMMARY:
TQD3606 is a fixed-dose combination of meropenem and avibatam. This study is a phase I clinical study to evaluate the safety, tolerability and pharmacokinetic characteristics of TQD3606 injection in a single center, randomized, double-blind, placebo-controlled, single and multiple administration in healthy subjects, and to explore the excretion of TQD3606 in urine. To evaluate the tolerability and safety of injectable TQD3606 after single and multiple dosing in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1 Signed the informed consent before the test and fully understood the test content, process and possible adverse reactions;
* 2 Able to complete the research according to the requirements of the test plan;
* 3 Subjects aged between 18 and 55 (including 18 and 55);
* 4 Body mass index (BMI) ≥ 18 and ≤ 28kg/m2, with male weight ≥ 50 kg and female weight ≥ 45 kg;
* 5 Health status: No mental disorders, no history of cardiovascular system, nervous system, respiratory system, digestive system, urinary system, endocrine system and metabolic abnormalities;
* 6 Subjects had no pregnancy plan and voluntarily used effective contraceptive measures for at least 6 months from 2 weeks before self-medication to the last use of study medication.

Exclusion Criteria:

* 1 Previous neuropsychiatric system, respiratory system, cardiovascular system, digestive system, hemolymph system, liver and kidney dysfunction, endocrine system, musculoskeletal system disease or other diseases, and the investigator judged that the previous history may affect drug metabolism or safety;
* 2 Known allergic history to meropenem or avitabtam, known history of anaphylactic shock to penicillin, cephalosporins, carbapenems and other β -lactam antibiotics or other severe allergic reactions (such as bullous epidermolysis atrophic dermatitis, exudative dermatitis);
* 3 Allergic constitution, including allergy to food and other drugs;
* 4 Persons with a history of epilepsy or central nervous system dysfunction;
* 5 Those with definite chronic headache or chronic diarrhea in the past;
* 6 Changes in QT interval or QT Corrected (QTc) > 450ms were considered clinically significant by researchers;
* 7 The creatinine clearance rate was less than 50ml/min;
* 8 Taking any prescription, over-the-counter, vitamin products or herbal medicine within 2 weeks prior to screening;
* 9 Abnormal and clinically significant laboratory tests during screening period;
* 10 Blood donation or significant blood loss within 3 months prior to taking the study drug (>450 ml);
* 11 Participated in any drug clinical trials within 3 months prior to taking the study drug;
* 12 Heavy smokers (5 cigarettes or more per day) within 3 months prior to screening;
* 13 Have a history of drug and/or alcohol abuse (14 units of alcohol per week: 1 unit =360mL beer or 45mL 40% spirits or 150mL wine);
* 14 Urine drug test positive or have a history of drug abuse or drug use in the past five years;
* 15 Unable to tolerate venipuncture blood collection or poor vascular condition;
* 16 Have taken a special diet (including dragon fruit, mango, grapefruit, grapefruit juice and/or xanthine diet) within 2 weeks prior to the trial;
* 17 Consuming chocolate, caffeinated coffee or tea within 48 hours before the trial;
* 18 Have taken any alcoholic food or beverage within 48 hours prior to the test;
* 19 The subject cannot complete the test due to personal reasons;
* 20 Conditions considered unsuitable for inclusion by other researchers.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Concentration (Cmax) | 1 hour before administration，to 24 hours after administration.
  Maximum Concentration
Area under the plasma concentration-time curve from initial dosing to 24 hours (AUC0-24) | 1 hour before administration，to 24 hours after administration.
  Area under the plasma concentration-time curve from initial dosing to 24 hours

SECONDARY OUTCOMES:
Time to maximum concentration following drug administration (Tmax) | 1 hour before administration，to 24 hours after administration.
  Time to maximum concentration following drug administration
Apparent terminal elimination half-life following drug administration (t1/2) | 1 hour before administration，to 24 hours after administration.
  Apparent terminal elimination half-life following drug administration
Area under plasma concentration-time curve from first dosing to last measurable concentration point (AUC0-t) | 1 hour before administration，to 24 hours after administration.
  Area under plasma concentration-time curve from first dosing to last measurable concentration point
The amount of drug excreted through urine 24 hours after administration (Ae0-24) | 1 hour before administration，to 24 hours after administration.
  The amount of drug excreted through urine 24 hours after administration
Cumulative excretion rate of drugs through urine | 1 hour before administration，to 24 hours after administration.
  Cumulative excretion rate of drugs through urine
The total clearance (CLt) The total clearance (CLt) | 1 hour before administration，to 24 hours after administration.
  The total clearance
Renal clearance (CLr) | 1 hour before administration，to 24 hours after administration.
  Renal clearance
Elimination rate constant(λz) | 1 hour before administration，to 24 hours after administration.
  Elimination rate constant
Apparent volume of distribution (Vd/F) | 1 hour before administration，to 24 hours after administration.
  Apparent volume of distribution
Mean residence time (MRT) | 1 hour before administration，to 24 hours after administration.
  Mean residence time
Valley concentration (Cmin,ss) | Within 60 minutes before 8th to 10th administration and 24 hours after 10th administration
  Valley concentration
Accumulation index | Within 60 minutes before 8th to 10th administration and 24 hours after 10th administration
  Accumulation index
Adverse event rate | Baseline up to 24 hours after administration
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Baseline up to 24 hours after administration
  Monitor the safety indicators of subjects during the trial
Body temperature | 1 hour before administration and 24 hours after administration
  Monitor the safety indicators of subjects during the trial
Pulse | 1 hour before administration and 24 hours after administration
  Monitor the safety indicators of subjects during the trial
Systolic and diastolic blood pressure | 1 hour before administration and 24 hours after administration
  Monitor the safety indicators of subjects during the trial
Number of participants with abnormal laboratory test results | Baseline up to 24 hours after administration
  Monitor the safety indicators of subjects during the trial

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun, Jilin, China